CLINICAL TRIAL: NCT06293573
Title: Comparative Effectiveness of Whole- Body Vibration and Aerobic Training Among Egyptian Elderly With Sarcopenia
Brief Title: Whole- Body Vibration Among Egyptian Elderly With Sarcopenia
Acronym: WBV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hussien Abdelmotaal Ali Elkadi, Assistant ecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/005031
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Elderly; Performance; Whole body vibration; Aerobic exercises
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be assigned randomly into three groups of equal number (study group A, study group B, and group C) the randomization will be performed by computerized randomization. Assessors will be blinded to the groups of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- whole body vibration group (Experimental): Group A (Study group): Will receive whole body vibration exercises with conventional progressive resistance exercises and diet modification life style
  Interventions: Device: Whole-body vibration; Other: resistance exercises
- aerobic exercise group (Experimental): Group B (Study group): Will receive aerobic exercises training with conventional progressive resistance exercises and diet modification life style.
  Interventions: Other: aerobic exercises; Other: resistance exercises
- conventional resistance exercise group (Active Comparator): Group C (Control Group): will receive conventional progressive resistance exercises and diet modification life style
  Interventions: Other: resistance exercises

INTERVENTIONS:
Device: Whole-body vibration — GROUP A : will receive whole body vibration exercises combined with resistance exercises
  Other Names: aerobic exercises - resistance exercises -life style
  Arms: whole body vibration group
Other: aerobic exercises — Group B will receive aerobic exercises training combined with progressive resistance exercises with diet modification life style.
  Arms: aerobic exercise group
Other: resistance exercises — Group c: will receive progressive resistance exercises with diet modification life style.

SUMMARY:
To investigate and compare between the effectiveness of whole body vibration and aerobic training exercises in management of sarcopenia, muscle mass, physical performance and muscle strength in elderly.

DETAILED DESCRIPTION:
Participants will be assigned randomly into two groups of equal number (study group A and study group B ) the randomization will be performed by computerized randomization. Assessors will be blinded to the groups of the subjects.

c- Subject selection 84 patients with sarcopenia will participate in this study and will be divided randomly into three equal groups with 28 participants in each group.

d- Groups: Group A (Study group): Will receive whole body vibration exercises with conventional progressive resistance exercises and diet modification life style Group B (Study group): Will receive aerobic exercises training with conventional progressive resistance exercises and diet modification life style.

Group C (Control Group): will receive conventional progressive resistance exercises and diet modification life style.

During the study, the participants will receive study information form, instructions and signed the consent form.

ELIGIBILITY:
Inclusion Criteria:

1. patients age older than 60 years
2. patients with Skeletal muscle index (SMI) below 8.87 kg/m2 and 6.42 kg/m2 in males and females, respectively.
3. patients with hand grip strength below < 27 kg in men and < 16 kg in women.
4. patients with no regular exercise habit for more than 3 months .
5. patients with gait speed > 0.8 m/s.
6. patients with proper conscious and cognition that will be detected by using Mini Mental State Examination(scores > 21).

   -

Exclusion Criteria:

acute injury. 2- severe heart diseases. 3- pacemaker. 4-history of orthopedic surgery of the lower limbs and/or fracture less than 1 year earlier.

.5 - inability to walk without assistance. 6-neurological diseases or acute conditions that would interfere with testing and training.

7-patients with improper conscious and cognition that will be detected by using Mini Mental State Examination(scores < 21).

8- patients who cannot exercise at all due to conditions like deep vein thrombosis or blood clotting issues.

9- patients with severe illnesses that influence assessments and interventions, such as those with disabilities or musculoskeletal conditions (such as fracture, dislocation, osteoporosis, and rheumatoid arthritis).

10- People with major spinal conditions or surgical histories, such as cauda equina syndrome, tumor, vertebral fracture, inflammatory joint disease, spondylolisthesis, and ankylosing spondylitis.

Every participant will get a primary checkup to get a full picture of their health, find out if there are any restrictions, and decide whether they can take part in the study.

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Mass | Muscle mass will be investigated at baseline and after the treatment period of 12 weeks.
  Outcome measures included:
  • Skeletal muscle mass (SMM): will be measured by Bioimpedance analysis using body composition analyzer (InBody Dial H 20b).
muscle strength | Muscle strength will be investigated at baseline and after the treatment period of 12 weeks.
  will be measured by using calibrated handheld dynamometer (CAMRY EH101).
timed Up and Go Test (TUG) | Timed Up and Go Test will be investigated at baseline and after the treatment period of 12 weeks.
  The TUG test evaluates physical function, individuals will be asked to rise from a standard chair, walk to a marker 3 m away from the chair, turn around, walk back, and sit down again.
Gait Speed test | Gait speed test will be investigated at baseline and after the treatment period of 12 weeks.
  The 4-m usual walking speed test, which measures speed either manually ,with a stopwatch or instrumentally, with an electronic device, to measure gait timing.
400 m Walking Test | 400 m Walking Test will be investigated at baseline and after the treatment period of 12 weeks.
  The 400-meters walk test evaluates a person's stamina and ability to walk. Participants in this test are required to run 20 laps of 20 meters, each lap as quickly as they can, and are permitted up to two rest breaks throughout the test.
Six minute walk test (6MWT) | Six Minutes Walk Test will be investigated at baseline and after the treatment period of 12 weeks.
  6MWT is used to measure a patient's exercise tolerance. Also it is used to assess aerobic capacity and endurance. Patient is asked to walk at his normal pace for six minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Embaby, phD, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt